CLINICAL TRIAL: NCT06131723
Title: UCLA Health Patient Health Tickler Email
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Richard K. Leuchter, MD, Clinical Instructor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AWVinitial
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Health Maintenance
Keywords: primary care; digital outreach

STUDY DESIGN:
Intervention Model Description: Parallel-arm control trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Standard tickler email (No Intervention): Eligible, assigned participants will receive the current standard email notification (i.e., "control tickler") from UCLA Health, informing patients that they have received a new message in their MyChart patient portal account, and containing links to their portal account.
- Arm 2: Enhanced tickler email (Experimental): Eligible, assigned participants will receive a behaviorally informed email notification (i.e., "enhanced tickler"), coming from their PCP's office, informing patients that they are due for an important medical exam, and containing a direct link to the MAP Letter on their patient portal account.
  Interventions: Behavioral: Behaviorally informed tickler email

INTERVENTIONS:
Behavioral: Behaviorally informed tickler email — The email notification from patients' PCP office will inform patients that a new review of their records shows they are due for an important medical exam. This intervention harnesses behavioral principles related to importance (medical exam described as important), personalization (records described as belonging to participants), urgency (participants are asked to sign in and make the recommended appointment as soon as possible), timeliness (participants are told that there has been a new review of their records), source effects and accountability (participants are told that a message from their PCP's office is waiting for their response). To make it easier for patients to find and review the MAP letter, the email also contains a link that directs patients to the MAP letter on their patient portal.
  Arms: Arm 2: Enhanced tickler email

SUMMARY:
This is a prospective clinical trial evaluating how a behaviorally-informed outreach email notification impacts patient engagement with primary care. This trial is being implemented in conjunction with UCLA Health's larger quality improvement initiative (the My Action Plan Quality Improvement Initiative) in order to improve primary care preventive measure completion rates.

The main question it aims to answer is if sending an enhanced email notification (i.e., enhanced tickler email) to identified UCLA Health primary care patients increases their engagement with primary care.

Participants will be assigned to either a control (standard tickler email) or treatment (enhanced tickler email) condition, based on whether their birth date ends in an odd or even number. Researchers will compare control and treatment groups to see if and how they differ in pre-defined outcome measures.

DETAILED DESCRIPTION:
Health maintenance measures have been shown to be critical in early detection, secondary prevention, and early management of numerous medical conditions--from diabetes to various cancers. The standardization of these health maintenance measures has resulted in major improvements in population health. Despite the importance of these primary care tests and screenings, many patients are overdue for these tests.

Given this healthcare gap, it is critical to investigate more effective strategies to communicate to patients about health maintenance measures they need to complete. This study aims to evaluate the effectiveness of a behaviorally-informed outreach email message. The investigators intend to launch the study as a part of UCLA Health's My Action Plan initiative, a UCLA Health primary care outreach quality improvement initiative aimed at encouraging patients to complete their overdue health maintenance measures.

Specifically, the My Action Plan (MAP) initiative is an outreach effort targeting primary care patients at UCLA Health who have outstanding, clinically indicated primary care preventative care gaps (e.g., overdue colorectal cancer screening, outstanding diabetes tests). At the beginning of the month following their birth month, patients with at least one of these open care gaps receive a MAP Letter in the form of a patient portal message. The MAP Letter contains a personalized list of outstanding preventive care items and actionable steps to complete the items. When the MAP Letter is received in the patient portal, it triggers an email "tickler" that is sent to patients' personal email address to notify them of the patient portal message.

At the beginning of each month, patients who are due to receive a MAP Letter will be assigned to receive either the current standard email tickler used by UCLA Health (control tickler) or a behaviorally-informed email tickler (enhanced tickler), based on whether their birth date ends in an odd or even number. The control email will notify them that they have a new message posted in their MyChart patient portal account, and prompt them to sign in to read it. The behaviorally-informed email will directly notify them that they are due for an important medical exam and prompt them to sign in to their MyChart patient portal account to schedule their recommended appointment; this message will be signed by their primary care doctor's office. In each month, emails will go out to all eligible patients in both conditions at the same time.

Both email notifications will contain links to the patient's MyChart portal account. The control tickler will link patients to their MyChart patient portal home page (standard procedure for email ticklers), whereas the enhanced tickler will link patients directly to the MAP Letter.

The investigators plan to run this clinical trial for 18 months.

By studying whether patients review the MAP letter and whether or not the engagement translates into completing health maintenance measures, the proposed study will provide insightful information on how health systems could optimize electronic patient outreach.

Analysis Plan:

* The investigators will utilize patient-level ordinary least squares (OLS) estimation, with statistical inferences based on model-robust standard errors. The primary model term will be an indicator variable for arm assignment.
* The analysis will control for sex, age, race/ethnicity, indicators for screenings/tests that patients are due for (which are marked on their MAP letter), and whether patients have upcoming primary care appointments at the time of MAP outreach. Missing covariate values will be handled by including 'unknown' indicators, along with mean imputation for quantitative covariates.
* The primary analyses will include patients who were contacted for the first time during our intervention period. For patients who reappear in the program between November 2024 and May 2025, the investigators will explore the effect of the second exposure to the redesigned tickler email within this subsample. Retargeting may be influenced by participants' original assignment to the control or treatment condition. For example, patients originally assigned to the enhanced tickler email condition may be more likely to close their care gap during the first exposure, reducing the likelihood of being retargeted in the second year. To address this potential endogeneity, the investigators will assess the balance between the control and treatment groups within the retargeted sample.
* Exploratory analyses will investigate heterogeneous treatment effects by patients' baseline motivation (i.e., the extent to which patients seem to have an intention to get the screenings/tests), which will be proxied by each patient's history of screenings/tests. Specifically, the investigators will calculate, among all the screenings/tests that are included in the My Action Plan Initiative and that a patient was due for in the past few years prior to the MAP outreach (the investigators aim for 10 years, but the exact time window is based on data availability), what percentage was completed by the patient (as far as UCLA Health could tell). A higher percentage indicates a higher baseline motivation to complete the screenings/tests patients are due for.
* The investigators will explore whether the difference between conditions is moderated by how frequently patients have seen their PCP in the past few years prior to the MAP outreach (the investigators target 3 years, but the exact time window is based on data availability).
* Additionally, the investigators will investigate whether the translation of engagement with the MAP Letter to actual appointment scheduling and screening/test completion (defined later in the secondary outcome section) depends on whether patients face structural barriers to get screenings/tests. The investigators will explore proxies including socioeconomic factors at the zipcode level (social vulnerability, income), insurance type, and distance from UCLA Health clinics (as a proxy for accessibility to healthcare).

ELIGIBILITY:
Inclusion Criteria:

1. Empaneled to UCLA Health DOM Primary Care
2. Has at least one overdue health maintenance measure that the My Action Plan initiative focuses on
3. Has an active MyChart status

Exclusion Criteria:

1. Under the age of 18
2. Deceased
3. In hospice
4. Has opted out of electronic communication (bulk messages, email, and/or text)
5. For the final analysis, the investigators will further exclude patients who have scheduled appointments for all screenings/tests or completed all screenings/tests prior to the date when they are supposed to receive the email notification, as well as patients who use proxies (e.g., family members who receive the email tickler on their behalf) given that all proxies are assigned to receive a standard tickler email.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81000 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
MAP Letter opened | From email notification outreach until 9 a.m. the next day before an automatic text reminder is sent to every participant, and 7 days after getting the outreach email notification
  Percentage of participants across the different arms who open their My Action Plan Letter on the MyChart patient portal

SECONDARY OUTCOMES:
Signing in to their MyChart patient portal | From email notification outreach until 9 a.m. the next day before an automatic text reminder is sent to every participant, and 7 days after getting the outreach email notification
  Percentage of participants across the different arms who sign in to their MyChart patient portal (irrespective of opening the MAP letter)
Visiting the appointment scheduling page | From email notification outreach until 9 a.m. the next day before an automatic text reminder is sent to every participant, and 7 days after getting the outreach email notification
  Percentage of participants across the different arms who visit the appointment scheduling page in their MyChart patient portal
Taking action for at least one overdue screening/test | From email notification outreach until 9 a.m. the next day before an automatic text reminder is sent to every participant, and 7 days after getting the outreach email notification
  Percentage of participants who schedule an appointment for at least one overdue screening/test or start the online tool for colorectal cancer screening (which is designed to help patients pick the screening modality and is the action item on MAP Letter for patients due for colorectal cancer screening).
Completing at least one screening/test | 6 months after getting the outreach email notification
  Percentage of participants who complete at least one screening/test

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health Department of Medicine, Quality Office, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make any individual participant data available.